CLINICAL TRIAL: NCT05898022
Title: Pragmatic Research on Diuretic Management in Early Bronchopulmonary Dysplasia (PRIMED) Pilot Study
Brief Title: Pragmatic Research on Diuretic Management in Early BPD Pilot
Acronym: PRIMED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rainbow Babies and Children's Hospital (Other); Emory University (Other); RTI International (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Heather Kaplan, Professor of Pediatrics, Children's Hospital Medical Center, Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0120; R34HL158586-01A1 (NIH)
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: furosemide; ventilator-induced lung injury; lung injury; lung diseases; respiratory tract diseases; infant; premature diseases; newborn; diseases; diuretics
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Ventilator-Induced Lung Injury; Lung Injury; Lung Diseases; Respiratory Tract Diseases; Disease | interventions — Furosemide

STUDY DESIGN:
Intervention Model Description: The proposed pilot, feasibility study will enroll patients in a series of N-of-1 trials. Each individual N-of-1 trial will have 2 blocks. In each block patients will crossover between furosemide (plus potassium chloride) for 4 days and placebo (plus placebo electrolyte solution) for 4 days. Each patient will have 8 days of total exposure to furosemide over the 16-day N-of-1 trial.
Masking Description: Participant, care provider, investigator, outcomes assessor learn the order of furosemide and placebo administration at the end of their N-of-1 trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- N-of-1 Trial (Other): Each individual N-of-1 trial will have 2 blocks. In each block patients will crossover between furosemide (plus potassium chloride) for 4 days and placebo (plus placebo electrolyte solution) for 4 days. The total arm length (length of the N-of-1 Trial/Crossover) is 16 days. Patients may receive furosemide (plus potassium chloride) and placebo (plus placebo electrolyte solution) in one of four different treatment order sequences, however, treatment order will not be analyzed for the primary outcomes of feasibility/responder status.
  Interventions: Drug: Furosemide (plus potassium chloride); Drug: Placebo (plus placebo electrolyte solution)

INTERVENTIONS:
Drug: Furosemide (plus potassium chloride) — Furosemide is a loop diuretic that inhibits the reabsorption of sodium and chloride in the proximal and distal tubules as well as the loop of Henle. Participants will receive 2 mg/kg enteral furosemide daily during treatment periods when they receive study drug. To prevent hypokalemia and hypochloremia associated with furosemide use, participants will also receive 1 mg/kg of potassium chloride enterally twice per day when receiving furosemide. Each patient will have 8 days of total exposure to furosemide over the 16-day N-of-1 trial.
Drug: Placebo (plus placebo electrolyte solution) — During treatment periods when participants receive placebo, they will receive a volume of sterile water equivalent to the study drug dose. Participants will also receive a placebo electrolyte solution equivalent to the volume of potassium chloride that would be given.

SUMMARY:
Babies who are born prematurely often develop a chronic lung disease called bronchopulmonary dysplasia (BPD). BPD puts babies at higher risk for problems with growth and development. Diuretics, such as furosemide, are frequently used in the management of early BPD). Many clinicians use informal trials of therapy to see if a baby responds to diuretics in the short-term before starting chronic diuretic therapy. Despite frequent use of diuretics, it is unclear how many babies truly respond to therapy and if there are long-term benefits of diuretic treatment. Designing research studies to figure this out has been challenging. The Pragmatic Research on Diuretic Management in Early BPD (PRIMED) study is a feasibility pilot study to help us get information to design a larger trial of diuretic management for BPD. Key questions this study will answer include: (1) Can we use an N-of-1 trial to determine whether a particular baby responds to furosemide? In an N-of-1 trial, a baby is switched between furosemide and placebo to compare that particular infant's response on and off diuretics. It is a more rigorous approach to the informal trials of therapy that are often conducted in clinical care. We hope to learn how many babies have a short-term response to furosemide ("responders"); (2) how many babies will still be on respiratory support at the end of the N-of-1 trial? This will help us determine how many patients would be eligible to randomize to chronic diuretic therapy in the second phase of the larger trail, and (3) if a baby is identified as a short-term responder, how many parents and physicians would be willing to randomize the baby to chronic diuretics (3 months) versus placebo in the longer trial?

ELIGIBILITY:
Inclusion Criteria:

1. <28 weeks gestation at birth
2. Post-Menstrual Age (PMA) of 29-32 weeks gestation
3. Requiring invasive positive pressure respiratory support or NIPPV/NIMV and FiO2 ≥ 25% or requiring non-invasive positive pressure respiratory support (NCPAP≥ 5 cm H20, BiPhasic CPAP) and FiO2 ≥ 30%.
4. Receiving enteral feedings of 120 mL/kg/day or greater
5. Expected to be hospitalized for at least 28 days after enrollment

Exclusion Criteria:

1. Major congenital anomalies (e.g., known renal anomalies, congenital heart disease, congenital diaphragmatic hernia, or chromosomal anomalies)
2. In infants who had electrolyte testing in the week prior to enrollment, those with a serum creatinine > 1.7 mg/dL, BUN >50 mg/dL, Na <125 mmoL/L, K ≤ 2.5 mmol/L, or Ca ≤ 6 mg/dL. Not having electrolyte testing in the week prior to enrollment is not an exclusion criterion.
3. Current treatment with Dexamethasone or hydrocortisone for respiratory failure. Treatment with chronic steroids for history of adrenal insufficiency or cardiovascular instability is not an exclusion criterion.
4. Treatment with any longer-acting diuretic (e.g., chlorothiazide, hydrochlorothiazide, acetazolamide) within 5 days of enrollment where exposure may result in carryover effects that confound the N-of-1 trial
5. Active order for standing, regularly scheduled diuretics (e.g., chronic diuretics)
6. Non-English speaking
7. Current treatment with ibuprofen or indocin

Ages: 2 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Percent of enrolled infants who completed the full N-of-1 trial, remain on respiratory support at the conclusion of the N-of-1 trial, and were identified as a responder | 23 Days
Percent of providers willing to support randomizing a responder infant | 30 Days

SECONDARY OUTCOMES:
Percent of enrolled infants completing full N-of-1 trial and identified as responder | 23 days
Percent of enrolled infants completing full N-of-1 trial | 23 days
Percent of enrolled infants on respiratory support at the conclusion of the N-of-1 trial | 23 days
Percent of parents willing to randomize responder infant | 30 days
Rate of chronic diuretic use among responders (and non-responders) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Heather Kaplan, MD, MSCE, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Anna Maria Hibbs, MD, MSCE, Principal Investigator — 1. Rainbow Babies and Children's Hospital
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - RTI International, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No